CLINICAL TRIAL: NCT02766842
Title: Evaluation of a New EUS Guided Biopsy Needle (SharkCore) Comparing to Standard EUS Needle (ProCore): A Prospective Randomized, Controlled Multicenter Study
Brief Title: Evaluation of a New EUS Guided Biopsy Needle (SharkCore) Comparing to Standard EUS Needle (ProCore)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason was the fact that the ProCore needle was removed from clinical use
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Mouen Khashab, Associate professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00095614
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Mesenchymal Tumor; Autoimmune Pancreatitis; Lymphoma; Solid Tumors
Keywords: SharkCore; ProCore
MeSH Terms: conditions — Autoimmune Pancreatitis; Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-FNB with ProCore needle (Active Comparator): General anesthesia or conscious sedation will be started and an upper endoscopic ultrasound will be inserted into the participants mouth and advanced to the site of the lesion. The lesion will be punctured by the ProCore needle, then the stylet is completely removed, and negative suction pressure is applied using a 10 ml syringe for 30 seconds while the needle is stationary with the target. Then, the needle is moved back and forth several times within the target, utilizing the fanning technique. Finally, suction is released by closing the lock of the syringe and the needle is removed.
  Interventions: Procedure: EUS-FNB with ProCore needle; Device: ProCore needle
- EUS-FNB with SharkCore needle (Active Comparator): The procedure will be done in the same manner with same endoscopic technique and method of tissue procurement. The only difference will be using the SharkCore needle to acquire tissue.
  Interventions: Procedure: EUS-FNB with SharkCore needle; Device: SharkCore needle

INTERVENTIONS:
Procedure: EUS-FNB with ProCore needle — The use of the standard ProCore needle to acquire diagnostic tissue
  Arms: EUS-FNB with ProCore needle
Procedure: EUS-FNB with SharkCore needle — The use of new SharkCore needle to acquire diagnostic tissue
  Arms: EUS-FNB with SharkCore needle
Device: ProCore needle — This is the standard needle used currently to procure tissue from lesions under endoscopic ultrasound guidance
  Arms: EUS-FNB with ProCore needle
Device: SharkCore needle — This is the new FDA approved needle for tissue procurement under endoscopic ultrasound guidance.
  Arms: EUS-FNB with SharkCore needle

SUMMARY:
Diagnosis of lesions of pancreas, the upper gastrointestinal tract, as well as adjacent structures, such as lymph nodes, is still showing advancements especially with the increased use of endoscopic ultrasound. Endoscopic ultrasound-guided fine needle aspiration and fine needle biopsy (EUS-FNA/FNB) have become mainstay diagnostic techniques for these lesions. The purpose of the study is to compare between the currently used, ProCore needles and the new biopsy needle, SharkCore, for the histological diagnosis and evaluation of lesions.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided fine needle aspiration and fine needle biopsy (EUS-FNA/FNB) have become mainstay diagnostic techniques for the diagnosis and evaluation of lesions of the pancreas, the upper gastrointestinal tract, as well as adjacent structures, including lymph nodes. Cytology specimens provided from FNA cannot fully characterize certain neoplasms such as lymphomas or mesenchymal tumors. Core biopsy specimens for histological examinations are needed to provide accurate diagnoses.

ProCore needles (ProCore, Wilson-Cook Medical Inc. Winston-Salem, NC) were designed to obtain histological and cytological samples. Studies comparing ProCore needles with standard FNA needles showed no significant difference in diagnostic accuracy, histological core tissue procurement or mean number of passes.

To overcome the above mentioned limitations (mainly suboptimal core tissue procurement rates), a new novel SharkCore needle (Beacon Endoscopic, Newton, MA, USA) has been designed and approved for clinical human use by the FDA.

The objective of the study is to compare the new EUS guided histology biopsy needle SharkCore to the currently used EUS histology needle, ProCore, for the histological diagnosis and evaluation of lesions.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 18 years of age referred for EUS

Lesions requiring histologic diagnosis:

* Mesenchymal tumors
* Autoimmune pancreatitis
* Granulomatous disease
* Indeterminate hepatitis
* Confirmatory immunochemistry to establish a diagnosis (i.e. pancreatic neuroendocrine tumor)
* Lymphoma
* Solid tumors
* Previously non-diagnostic FNA

Exclusion Criteria:

* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Uncooperative patients
* Pregnant women (women of childbearing age will undergo urine pregnancy testing, which is routine for all endoscopic procedures)
* Refusal to consent form
* Cystic lesions
* Inaccessible lesions to EUS (proximal to sigmoid colon or distal to second duodenum)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of needle as assessed by diagnostic yield of needle and final diagnosis method | Up to 1 month
  The final diagnosis of tissue from needle will be compared to the final diagnosis reached either by surgical removal of mass or other method of biopsy

SECONDARY OUTCOMES:
Number of passes to procure core tissue from needle | During procedure
  The number of passes needed to acquire core tissue as assessed by the pathologist in the room.
Safety of tissue procurement by needle | Up to 1 year
  All complications related to needle used will be recorded with a preset questionnaire to measure the frequency of complications related to needle used.
Procedure time | During procedure
  Time required to acquire tissue using each needle will be recorded from time of needle insertion to time of core tissue procurement as per pathologist.

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided